CLINICAL TRIAL: NCT06046352
Title: Symptom Burden Guiding Invasive Electrophysiological Study in Paroxysmal Supraventricular Tachycardia
Acronym: BELIEVE-SVT
Status: Completed | Type: Observational
Sponsor: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor
Other Study IDs: 19/562
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Supraventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Supraventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Non-documented, clinically-suspected PSVT
  Interventions: Procedure: Electrophysiological study (and ablation when appropriate)

INTERVENTIONS:
Procedure: Electrophysiological study (and ablation when appropriate) — Electrophysiological study (and ablation when appropriate)

SUMMARY:
BELIEVE-SVT is a European multi-centre, retrospective registry in tertiary hospitals performing electrophysiological study in patients with palpitations considered clinically suggestive of paroxysmal supraventricular tachycardia by a cardiologist and without electrocardiographic documentation of tachycardia or preexcitation. Clinical characteristics, results of electrophysiological study and ablation, complications, and clinical outcomes during follow-up will be analysed.

DETAILED DESCRIPTION:
The "Symptom Burden As Guiding Principle For Invasive Electrophysiological Study In Paroxysmal Supraventricular Tachycardia (Believe-SVT)" study was a multi-centre, retrospective, observational registry carried out in tertiary European hospitals. Inclusion criteria were: symptoms that were considered suggestive of paroxysmal supraventricular tachycardia by a cardiologist and/or cardiac electrophysiologist; absence of any sort of electrocardiographic tracing during episodes (including wearables and other single lead devices), and having undergone an electrophysiological study aimed at the diagnosis of paroxysmal supraventricular tachycardia.

ELIGIBILITY:
Inclusion criteria:

* Symptoms that were considered suggestive of paroxysmal supraventricular tachycardia by a cardiologist and/or cardiac electrophysiologist
* Absence of any sort of ECG tracing during episodes (including wearables and other single lead devices)

Exclusion criteria:

* Documentation of preexcitation
* Prior electrophysiological study aimed at the assessment of ventriculo-atrial conduction or induction of supraventricular tachycardias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with palpitations clinically suggestive of paroxysmal supraventricular tachycardia but no ECG documentation of tachycardia
Sampling Method: Non-Probability Sample
Enrollment: 711 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Electrophysiological study findings | 5 years
  Number of participants in whom paroxysmal supraventricular tachycardia or evidence of substrate enabling paroxysmal supraventricular tachycardia is observed in electrophysiological study

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rodriguez, MD PhD, Principal Investigator — University Hospital 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No